CLINICAL TRIAL: NCT00239473
Title: A Randomised, Double-Blind, Double-Dummy, Placebo- and Active-Controlled, Parallel Group Efficacy and Safety Comparison of 12-Week Treatment of Two Doses [5 μg (2 Actuations of 2.5 μg) and 10 μg (2 Actuations of 5 μg)] of Tiotropium Inhalation Solution Delivered by the Respimat Inhaler, Placebo and Ipratropium Bromide Inhalation Aerosol (MDI) in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: 12 Week Comparison of 5 Mcg and 10 Mcg of Tiotropium / Respimat, Placebo and Ipratropium MDI in COPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205.251
Record Dates: First submitted 2005-10-14; First posted 2005-10-17 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

INTERVENTIONS:
Device: 5 mcg once daily tiotropium inhalation solution delivered by the Respimat inhaler
Device: 10 mcg once daily tiotropium inhalation solution delivered by the Respimat inhaler

SUMMARY:
The primary objective was to compare the bronchodilator efficacy of two doses (5 mcg and 10 mcg) of tiotropium inhalation solution delivered by the Respimat inhaler once daily to placebo and to ipratropium bromide MDI four times daily in patients with COPD. The secondary objective was to compare the safety of tiotropium inhalation solution delivered by the Respimat to placebo and ipratropium bromide MDI.

ELIGIBILITY:
Outpatients of either sex, aged >/= 40 years with a diagnosis of COPD (FEV1 </= 60% predicted [ECCS criteria] and FEV1/FVC </= 70%)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 429
Dates: Start 2002-11; Primary Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Trough FEV1 response | after 12 weeks

SECONDARY OUTCOMES:
Trough FEV1 response | after 1, 4 and 8 weeks
Trough FVC response | after 1, 4, 8 and 12 weeks
FEV1 and FVC area under the curve (AUC)0-6h and peak response | after 0, 1, 4, 8 and 12 weeks
Individual FEV1 and FVC measurements | during 12 weeks
Onset and duration of therapeutic response and percentage of responders | after 0 and 12 weeks
Weekly mean pre-dose morning and evening PEFR (peak expiratory flow rate) | up to 12 weeks
Weekly mean number of occasions of rescue therapy used per day (PRN salbutamol) | up to 12 weeks
COPD symptom scores (wheezing, shortness of breath, coughing and tightness of chest) | up to 15 weeks
Physician's Global Evaluation | up to 15 weeks
Number of patients with at least one exacerbation of COPD | up to 15 weeks
Time to first exacerbation | up to 15 weeks
Number of exacerbations and exacerbation days | up to 15 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — Boehringer Ingelheim
Locations (38):
- Germany (17):
  - Boehringer Ingelheim Investigational Site, Berlin
  - MEDARS GmbH, Berlin
  - Boehringer Ingelheim Investigational Site, Bonn
  - Boehringer Ingelheim Investigational Site, Frankfurt am Main
  - Inamed Research GmbH & Co. KG, Gauting
  - Pneumologisches Forschungsinstitut GmbH, Großhansdorf
  - Pneumologisches Forschungsinstitut GmbH am Krankenhaus, Hamburg
  - Boehringer Ingelheim Investigational Site, Hanover
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - ClinPharm International GmbH & Co. KG, Leipzig
  - Neurologische Klinik der Otto-von-Guericke-Universität, Magdeburg
  - Johannes-Gutenberg-Universität Mainz, Mainz
  - Boehringer Ingelheim Investigational Site, Minden
  - Medizinische Klinik III, Moers
  - Boehringer Ingelheim Investigational Site, München
  - Abt. Lungen- und Bronchialheilkunde, Schmallenberg
  - Boehringer Ingelheim Investigational Site, Steinfurt
- Italy (9):
  - Ospedale Generale Provinciale Mazzoni, Ascoli Piceno
  - Dip. di Medicina Interna e Medicina Specialistica, Catania
  - U. O. di Fisiopatologia Respiratoria, Ferrara
  - Ospedale S. Martino, Genova
  - U. O. di Pneumologia e Servizio di Fisiopatologia Resp., Milan
  - IRCCS Policlinico San Matteo, Pavia
  - U. O. C di Pneumologia, Roma
  - Ospedale Silvestrini, San Sisto (pg)
  - U. O. di Pneumologia, Trieste
- South Africa (4):
  - Hydromed Hospital, Bloemfontein
  - UCT Lung Institute, Cape Town
  - 1 Military Hospital, Pretoria
  - Tygerberg Hospital, Tygerberg
- Switzerland (8):
  - Universitätskliniken Basel, Basel
  - Ospedale San Giovanni, Bellinzona
  - Boehringer Ingelheim Investigational Site, Davos
  - Boehringer Ingelheim Investigational Site, Laufen
  - Boehringer Ingelheim Investigational Site, Locarno
  - Ospedale Regionale, Lugano
  - Boehringer Ingelheim Investigational Site, Münchenstein
  - Kantonsspital St. Gallen, Sankt Gallen